CLINICAL TRIAL: NCT05537571
Title: A Multi-centre, Randomised, Double-blind, Placebo-controlled, Phase 2 Study to Investigate Efficacy, Safety and Tolerability of SLN360 in Participants With Elevated Lipoprotein(a) at High Risk of Atherosclerotic Cardiovascular Disease Events
Brief Title: Evaluate SLN360 in Participants With Elevated Lipoprotein(a) at High Risk of Atherosclerotic Cardiovascular Disease Events
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Silence Therapeutics plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLN360-002
Record Dates: First submitted 2022-09-06; First posted 2022-09-13 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Lipoprotein(a)
Keywords: Cardiovascular Diseases; Atherosclerosis; Lipoprotein(a)
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- SLN360 300 mg Q16W (Experimental): SLN360 300 mg administered subcutaneously at Weeks 0, 16 and 32 (Q16W)
  Interventions: Drug: SLN360
- SLN360 300 mg Q24W (Experimental): SLN360 300 mg administered subcutaneously at Weeks 0 and 24 (Q24W)
  Interventions: Drug: SLN360
- SLN360 450 mg Q24W (Experimental): SLN360 450 mg administered subcutaneously at Weeks 0 and 24 (Q24W)
  Interventions: Drug: SLN360
- Placebo Q16W (Placebo Comparator): Placebo administered subcutaneously at Weeks 0, 16 and 32 (Q16W)
  Interventions: Drug: Placebo
- Placebo Q24W (Placebo Comparator): Placebo administered subcutaneously at Weeks 0 and 24 (Q24W). This group was stratified so that half of participants were dosed to match the SLN360 300 mg Q24W group and half were dosed to match the SLN360 450 mg Q24W group (with respect to injected volume)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SLN360 — SLN360 is a double-stranded small interfering ribonucleic acid (siRNA) targeting LPA messenger RNA (mRNA)
  Other Names: Zerlasiran
  Arms: SLN360 300 mg Q16W; SLN360 300 mg Q24W; SLN360 450 mg Q24W
Drug: Placebo — Sodium chloride, solution for injection
  Arms: Placebo Q16W; Placebo Q24W

SUMMARY:
Phase 2 study to evaluate the efficacy, safety and tolerability of SLN360 administered subcutaneously (SC) compared with placebo in adult participants with elevated lipoprotein(a) at high risk of atherosclerotic cardiovascular disease events

ELIGIBILITY:
Inclusion Criteria:

* Lipoprotein(a) at screening equal to or greater than 125 nmol/L
* At high risk of ASCVD events
* A body mass index at screening in the range of 18.0 to 32.0 kg/m², inclusive

Exclusion Criteria:

* Renal dysfunction with estimated glomerular filtration rate less than 30 mL/min/1.73 m² at screening
* History or clinical evidence of hepatic dysfunction
* Malignancy within the 5 years before screening
* Fasting triglycerides >400 mg/dL (4.5 mmol/L) at screening
* Currently receiving or <12 weeks at Day 1 since receiving >200 mg/day niacin or niacin derivative drugs
* Treatment with lipid/lipoprotein apheresis within the 12 weeks before screening
* Any previous use of approved or experimental small interfering RNA (siRNA) therapy (e.g. inclisiran). NB: use of messenger RNA (mRNA) based vaccines for infectious diseases is permitted

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- Australia (3):
  - Royal Adelaide Hospital, Adelaide
  - Monash Health, Melbourne
  - Linear Clinical Research, Nedlands
- Czechia (4):
  - Medicus Services SRO, Brandýs nad Labem
  - Edumed s.r.o., Kardiologicka, endokrinologicka, diabetologicka a interni ambulance Nachod, Náchod
  - Pratia Pardubice a.s., Pardubice
  - Endokrinologie Cerny Most s.r.o., Prague
- Denmark (3):
  - Gentofte Hospital, Hellerup
  - Regionshospitalet Godstrup, Herning
  - Viborg Regional Hospital, Viborg
- Netherlands (5):
  - Academic Medical Center - Department of Vascular Medicine, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Bravis Ziekenhuis - Bergen op Zoom, Roosendaal
  - Universitair Medisch Centrum Utrecht, Utrecht
  - VieCuri Medisch Centrum, Venlo
- Slovakia (2):
  - Alian, s.r.o., Kardiologicka ambulancia, Bardejov
  - Kardiomed s.r.o., Lučenec
- South Africa (7):
  - Iatros International, Bloemfontein
  - Tiervlei Trial Centre (TTC), Cape Town
  - TREAD Research - Department of Cardiology, Cape Town
  - University of Cape Town - Lipid Laboratory, Cape Town
  - Paarl Research Centre, Paarl
  - Dr JM Engelbrecht Trial Site, Somerset West
  - Helderberg Research Institute, Somerset West
- United Kingdom (5):
  - Royal Sussex County Hospital, Brighton
  - Chelsea and Westminster Hospital, London
  - Panthera - London North, London
  - Panthera - Manchester, Rochdale
  - Panthera - Sheffield, Sheffield

REFERENCES:
- [Result] Nissen SE, Wang Q, Nicholls SJ, Navar AM, Ray KK, Schwartz GG, Szarek M, Stroes ESG, Troquay R, Dorresteijn JAN, Fok H, Rider DA, Romano S, Wolski K, Rambaran C. Zerlasiran-A Small-Interfering RNA Targeting Lipoprotein(a): A Phase 2 Randomized Clinical Trial. JAMA. 2024 Dec 17;332(23):1992-2002. doi: 10.1001/jama.2024.21957. PMID 39556769
- [Derived] Nicholls SJ. Therapeutic lowering of lipoprotein(a): implications for improving outcomes in patients with peripheral arterial disease. Curr Opin Lipidol. 2025 Oct 1;36(5):232-237. doi: 10.1097/MOL.0000000000001002. Epub 2025 Jul 21. PMID 40699211
- [Derived] Nicholls SJ, Nelson AJ, Michael LF. Oral agents for lowering lipoprotein(a). Curr Opin Lipidol. 2024 Dec 1;35(6):275-280. doi: 10.1097/MOL.0000000000000953. Epub 2024 Sep 25. PMID 39329200
- [Derived] Dimitriadis K, Theofilis P, Iliakis P, Pyrpyris N, Dri E, Sakalidis A, Soulaidopoulos S, Tsioufis P, Fragkoulis C, Chrysohoou C, Tsiachris D, Tsioufis K. Management of dyslipidemia in coronary artery disease: the present and the future. Coron Artery Dis. 2024 Sep 1;35(6):516-524. doi: 10.1097/MCA.0000000000001375. Epub 2024 Apr 29. PMID 38682459
- See also: PubMed Publication — http://www.ncbi.nlm.nih.gov/pubmed/39556769

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened from 05 December 2022, first randomised participant signed informed consent on 13 December 2022 and last participant was randomised 27 April 2023.
Pre-assignment Details: A total of 253 participants were screened for inclusion, 73 participants failed screening.
Period: Overall Study
Arm/Group | SLN360 300 mg Q16W | SLN360 300 mg Q24W | SLN360 450 mg Q24W | Placebo Q16W | Placebo Q24W
Started | 44 | 44 | 45 | 23 | 24
Completed | 39 | 43 | 44 | 23 | 23
Not Completed | 5 | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0
Not completed — Hepatitis A screening result | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline data are based on the set of unique participants who were randomised and treated. This excludes 2 participant numbers that enrolled but were not treated, due to hepatitis A screening results, but were later rescreened and re-randomised / treated.
Groups:
- Placebo Q16W: Placebo administered subcutaneously at Weeks 0, 16 and 32 (dosing every 16 weeks [Q16W])
  Placebo: Sodium chloride, solution for injection
- Placebo Q24W: Placebo administered subcutaneously at Weeks 0 and 24 (dosing every 24 weeks [Q24W]). This group was stratified so that half of participants were dosed to match the SLN360 300 mg Q24W group and half were dosed to match the SLN360 450 mg Q24W group (with respect to injected volume).
  Placebo: Sodium chloride, solution for injection
- Total: Total of all reporting groups
Arm/Group | SLN360 300 mg Q16W | SLN360 300 mg Q24W | SLN360 450 mg Q24W | Placebo Q16W | Placebo Q24W | Total
Number analyzed (Participants) | 42 | 44 | 45 | 23 | 24 | 178
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 23 | 22 | 12 | 15 | 91
  >=65 years | 23 | 21 | 23 | 11 | 9 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (9.81) | 64.5 (8.67) | 63.8 (10.23) | 65.0 (8.79) | 62.1 (9.43) | 63.7 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 11 | 5 | 6 | 46
  Male | 31 | 31 | 34 | 18 | 18 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 42 | 44 | 45 | 23 | 24 | 178
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 4 | 0 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 0 | 0 | 3
  White | 38 | 36 | 36 | 21 | 22 | 153
  More than one race | 2 | 5 | 3 | 2 | 1 | 13
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Netherlands | 13 | 15 | 16 | 8 | 8 | 60
  Czechia | 2 | 1 | 2 | 3 | 3 | 11
  Denmark | 7 | 9 | 3 | 3 | 3 | 25
  United Kingdom | 9 | 6 | 9 | 5 | 3 | 32
  South Africa | 6 | 8 | 9 | 3 | 3 | 29
  Slovakia | 2 | 0 | 3 | 0 | 0 | 5
  Australia | 3 | 5 | 3 | 1 | 4 | 16
Time from the initial date of elevated Lipoprotein(a) to randomisation date [Median (Inter-Quartile Range); unit: months] | 6.10 [1.30 to 12.10] | 5.45 [1.05 to 17.95] | 3.70 [1.30 to 11.50] | 3.60 [0.80 to 15.80] | 5.35 [1.20 to 28.70] | 4.45 [1.20 to 14.20]
Weight [Median (Inter-Quartile Range); unit: kilograms] | 84.15 [78.00 to 94.80] | 82.60 [73.65 to 95.70] | 80.20 [66.30 to 85.30] | 81.00 [66.20 to 91.20] | 84.10 [76.15 to 89.05] | 82.85 [72.20 to 91.10]
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m2] | 27.060 [25.080 to 29.750] | 28.240 [23.655 to 30.235] | 26.470 [24.540 to 28.440] | 26.930 [24.770 to 29.980] | 26.160 [25.105 to 27.920] | 26.905 [24.640 to 29.690]
Height [Median (Inter-Quartile Range); unit: centimetres] | 177.0 [170.0 to 182.0] | 175.0 [167.5 to 183.0] | 173.0 [164.0 to 180.0] | 170.0 [166.0 to 184.0] | 174.5 [171.5 to 183.5] | 175.0 [168.0 to 183.0]

OUTCOME MEASURES:

1. Primary Outcome: Time-averaged Percent Change In Lipoprotein(a) Molar Concentration From Baseline to Week 36
Description: Clinical trial results (relative to Day 1 pre-dose) was calculated for each participant by estimating the sum of the area under the curve with the linear trapezoidal method for all scheduled assessments from Week 4 to Week 36, inclusive, divided by the total time interval between the Week 4 and Week 36 assessments. Analysis of variance was used to test for differences between each active treatment group and the pooled placebo groups in the primary outcome measure. Time-averaged percent change in lipoprotein(a) to Week 36 was the dependent variable, and treatment group was included as the predictor variable. The least squares means, standard errors, and 2-sided 95% confidence intervals for each treatment group and for the pairwise comparisons between the SLN360 and placebo groups were estimated.
Time Frame: Week 36
Population: The pharmacodynamic population included all participants who received at least 1 dose of study drug and had evaluable pharmacodynamic data.
Measure: Least Squares Mean (Standard Error); unit: Percentage
Groups:
- Pooled Placebo: Pooled data from both placebo groups
  Placebo: Sodium chloride, solution for injection
Arm/Group | SLN360 300 mg Q16W | SLN360 300 mg Q24W | SLN360 450 mg Q24W | Pooled Placebo
Number analyzed (Participants) | 42 | 44 | 45 | 47
Percentage | -80.5 (1.99) | -79.1 (1.94) | -83.3 (1.92) | 2.3 (1.88)
Statistical Analysis 1: Comparison: SLN360 300 mg Q16W vs Pooled Placebo; Analysis of variance (ANOVA) was used to test for differences between each active treatment group and the pooled placebo groups in the primary outcome measure; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Final Values) = -82.8, 95% CI 2-sided [-88.19 to -77.39]
Statistical Analysis 2: Comparison: SLN360 300 mg Q24W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Final Values) = -81.3, 95% CI 2-sided [-86.68 to -76.0]
Statistical Analysis 3: Comparison: SLN360 450 mg Q24W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Final Values) = -85.6, 95% CI 2-sided [-90.88 to -80.26]

2. Secondary Outcome: Time-averaged Percent Change In Lipoprotein(a) Molar Concentration From Baseline to Week 48
Description: Time-averaged secondary endpoints were calculated and analysed using the same conventions as the primary endpoint.
Time Frame: Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | SLN360 300 mg Q16W | SLN360 300 mg Q24W | SLN360 450 mg Q24W | Pooled Placebo
Number analyzed (Participants) | 42 | 44 | 45 | 47
Percentage | -81.6 (2.05) | -77.2 (2.00) | -81.5 (1.98) | 1.5 (1.94)
Statistical Analysis 1: Comparison: SLN360 300 mg Q16W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Final Values) = -83.1, 95% CI 2-sided [-88.7 to -77.57]
Statistical Analysis 2: Comparison: SLN360 300 mg Q24W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Final Values) = -78.7, 95% CI 2-sided [-84.18 to -73.17]
Statistical Analysis 3: Comparison: SLN360 450 mg Q24W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Final Values) = -83.0, 95% CI 2-sided [-88.43 to -77.49]

3. Secondary Outcome: Time-averaged Percent Change In Lipoprotein(a) Molar Concentration From Baseline to Week 60
Description: Time-averaged secondary endpoints were calculated and analysed using the same conventions as the primary endpoint.
Time Frame: Week 60
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | SLN360 300 mg Q16W | SLN360 300 mg Q24W | SLN360 450 mg Q24W | Pooled Placebo
Number analyzed (Participants) | 42 | 44 | 45 | 47
Percentage | -78.0 (2.24) | -70.7 (2.19) | -76.0 (2.16) | 1.1 (2.11)
Statistical Analysis 1: Comparison: SLN360 300 mg Q16W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Final Values) = -79.2, 95% CI 2-sided [-85.25 to -73.1]
Statistical Analysis 2: Comparison: SLN360 300 mg Q24W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Final Values) = -71.8, 95% CI 2-sided [-77.81 to -65.8]
Statistical Analysis 3: Comparison: SLN360 450 mg Q24W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Final Values) = -77.1, 95% CI 2-sided [-83.09 to -71.15]

4. Secondary Outcome: Time-averaged Percent Change In Apolipoprotein B Concentration From Baseline to Week 36
Description: Time-averaged secondary endpoints were calculated and analysed using the same conventions as the primary endpoint.
Time Frame: Week 36
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | SLN360 300 mg Q16W | SLN360 300 mg Q24W | SLN360 450 mg Q24W | Pooled Placebo
Number analyzed (Participants) | 42 | 44 | 45 | 47
Percentage | -16.9 (1.93) | -13.5 (1.88) | -18.6 (1.86) | -3.6 (1.82)
Statistical Analysis 1: Comparison: SLN360 300 mg Q16W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Final Values) = -13.3, 95% CI 2-sided [-18.55 to -8.09]
Statistical Analysis 2: Comparison: SLN360 300 mg Q24W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0002, ANOVA; Mean Difference (Final Values) = -9.9, 95% CI 2-sided [-15.02 to -4.68]
Statistical Analysis 3: Comparison: SLN360 450 mg Q24W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Final Values) = -15.0, 95% CI 2-sided [-20.1 to -9.82]

5. Secondary Outcome: Time-averaged Percent Change In Apolipoprotein B Concentration From Baseline to Week 48
Description: Time-averaged secondary endpoints were calculated and analysed using the same conventions as the primary endpoint.
Time Frame: Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | SLN360 300 mg Q16W | SLN360 300 mg Q24W | SLN360 450 mg Q24W | Pooled Placebo
Number analyzed (Participants) | 42 | 44 | 45 | 47
Percentage | -16.4 (1.94) | -12.6 (1.90) | -18.0 (1.88) | -4.0 (1.83)
Statistical Analysis 1: Comparison: SLN360 300 mg Q16W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Final Values) = -12.3, 95% CI 2-sided [-17.62 to -7.08]
Statistical Analysis 2: Comparison: SLN360 300 mg Q24W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0013, ANOVA; Mean Difference (Final Values) = -8.6, 95% CI 2-sided [-13.85 to -3.44]
Statistical Analysis 3: Comparison: SLN360 450 mg Q24W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Final Values) = -14.0, 95% CI 2-sided [-19.2 to -8.84]

6. Secondary Outcome: Time-averaged Percent Change In Apolipoprotein B Concentration From Baseline to Week 60
Description: Time-averaged secondary endpoints were calculated and analysed using the same conventions as the primary endpoint.
Time Frame: Week 60
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | SLN360 300 mg Q16W | SLN360 300 mg Q24W | SLN360 450 mg Q24W | Pooled Placebo
Number analyzed (Participants) | 42 | 44 | 45 | 47
Percentage | -15.0 (2.04) | -10.9 (1.99) | -16.4 (1.97) | -3.8 (1.93)
Statistical Analysis 1: Comparison: SLN360 300 mg Q16W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Final Values) = -11.3, 95% CI 2-sided [-16.81 to -5.73]
Statistical Analysis 2: Comparison: SLN360 300 mg Q24W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0106, ANOVA; Mean Difference (Final Values) = -7.2, 95% CI 2-sided [-12.64 to -1.69]
Statistical Analysis 3: Comparison: SLN360 450 mg Q24W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANOVA; Mean Difference (Final Values) = -12.6, 95% CI 2-sided [-18.04 to -7.15]

7. Secondary Outcome: Time-averaged Percent Change In Low-density Lipoprotein Cholesterol Concentration From Baseline to Week 36
Description: Time-averaged secondary endpoints were calculated and analysed using the same conventions as the primary endpoint.
Time Frame: Week 36
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | SLN360 300 mg Q16W | SLN360 300 mg Q24W | SLN360 450 mg Q24W | Pooled Placebo
Number analyzed (Participants) | 42 | 44 | 45 | 47
Percentage | -22.3 (8.16) | -20.1 (7.98) | -15.5 (7.89) | 9.6 (7.72)
Statistical Analysis 1: Comparison: SLN360 300 mg Q16W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0051, ANOVA; Mean Difference (Final Values) = -31.9, 95% CI 2-sided [-54.07 to -9.72]
Statistical Analysis 2: Comparison: SLN360 300 mg Q24W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0081, ANOVA; Mean Difference (Final Values) = -29.7, 95% CI 2-sided [-51.62 to -7.81]
Statistical Analysis 3: Comparison: SLN360 450 mg Q24W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0241, ANOVA; Mean Difference (Final Values) = -25.1, 95% CI 2-sided [-46.89 to -3.33]

8. Secondary Outcome: Time-averaged Percent Change In Low-density Lipoprotein Cholesterol Concentration From Baseline to Week 48
Description: Time-averaged secondary endpoints were calculated and analysed using the same conventions as the primary endpoint.
Time Frame: Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | SLN360 300 mg Q16W | SLN360 300 mg Q24W | SLN360 450 mg Q24W | Pooled Placebo
Number analyzed (Participants) | 42 | 44 | 45 | 47
Percentage | -20.9 (7.01) | -18.5 (6.85) | -17.0 (6.78) | 8.9 (6.63)
Statistical Analysis 1: Comparison: SLN360 300 mg Q16W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0023, ANOVA; Mean Difference (Final Values) = -29.8, 95% CI 2-sided [-48.86 to -10.76]
Statistical Analysis 2: Comparison: SLN360 300 mg Q24W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0046, ANOVA; Mean Difference (Final Values) = -27.4, 95% CI 2-sided [-46.23 to -8.58]
Statistical Analysis 3: Comparison: SLN360 450 mg Q24W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0068, ANOVA; Mean Difference (Final Values) = -26.0, 95% CI 2-sided [-44.67 to -7.24]

9. Secondary Outcome: Time-averaged Percent Change In Low-density Lipoprotein Cholesterol Concentration From Baseline to Week 60
Description: Time-averaged secondary endpoints were calculated and analysed using the same conventions as the primary endpoint.
Time Frame: Week 60
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | SLN360 300 mg Q16W | SLN360 300 mg Q24W | SLN360 450 mg Q24W | Pooled Placebo
Number analyzed (Participants) | 42 | 44 | 45 | 47
Percentage | -19.3 (7.45) | -16.8 (7.28) | -14.7 (7.19) | 9.3 (7.04)
Statistical Analysis 1: Comparison: SLN360 300 mg Q16W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0057, ANOVA; Mean Difference (Final Values) = -28.7, 95% CI 2-sided [-48.91 to -8.46]
Statistical Analysis 2: Comparison: SLN360 300 mg Q24W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = -26.1, 95% CI 2-sided [-46.13 to -6.16]
Statistical Analysis 3: Comparison: SLN360 450 mg Q24W vs Pooled Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0179, ANOVA; Mean Difference (Final Values) = -24.1, 95% CI 2-sided [-43.93 to -4.2]

ADVERSE EVENTS:
Time Frame: 05 December 2022 (first participant screened) to 01 July 2024 (last participant last visit). Median duration of exposure was 24.43 weeks. Adverse event data were collected over the 60-week study period (95.6% of participants completed to Week 60).
Description: Serious treatment-emergent and non-serious treatment-emergent adverse events are summarised for the safety population: all participants who received at least 1 dose of study drug. Safety data were summarised by actual treatment received based on the safety population.
Groups:
- Placebo Q16W: Placebo administered subcutaneously at Weeks 0, 16 and 32 (dosing every 16 weeks [Q16W]).
  Placebo: Sodium chloride, solution for injection
Arm/Group | SLN360 300 mg Q16W | SLN360 300 mg Q24W | SLN360 450 mg Q24W | Placebo Q16W | Placebo Q24W
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/44 | 0/45 | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 6/42 | 2/44 | 5/45 | 1/23 | 3/24
Other Adverse Events (participants affected / at risk) | 42/42 | 43/44 | 42/45 | 18/23 | 22/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SLN360 300 mg Q16W (N=42) | SLN360 300 mg Q24W (N=44) | SLN360 450 mg Q24W (N=45) | Placebo Q16W (N=23) | Placebo Q24W (N=24)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute vestibular syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymph node tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SLN360 300 mg Q16W (N=42) | SLN360 300 mg Q24W (N=44) | SLN360 450 mg Q24W (N=45) | Placebo Q16W (N=23) | Placebo Q24W (N=24)
Procedural pain (Injury, poisoning and procedural complications) | 4 (8) | 1 (1) | 2 (4) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (2) | 2 (2) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3) | 4 (5) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 3 (5) | 6 (8) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Influenza-like illness (General disorders) | 2 (2) | 1 (1) | 7 (7) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 35 (71) | 36 (55) | 37 (109) | 2 (3) | 2 (2)
Malaise (General disorders) | 6 (8) | 0 (0) | 4 (5) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 4 (4) | 2 (2) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 7 (8) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 6 (7) | 4 (4) | 3 (3) | 4 (4)
Nasopharyngitis (Infections and infestations) | 3 (3) | 6 (8) | 6 (9) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 7 (8) | 5 (5) | 1 (1) | 3 (6)
Urinary tract infection (Infections and infestations) | 5 (6) | 1 (2) | 3 (4) | 3 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT05537571/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT05537571/SAP_001.pdf